CLINICAL TRIAL: NCT05108246
Title: Home-Based Dual-Task Training to Improve Function in Older Adults
Brief Title: Home-Based Dual-Task Training for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Nikhil Satchidanand, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004857; UL1TR001412 (NIH)
Record Dates: First submitted 2021-10-13; First posted 2021-11-04 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-Task Training (Experimental): Dual-Task Exercise
  Interventions: Behavioral: Dual-Task Exercise Training
- Control (No Intervention): No Exercise

INTERVENTIONS:
Behavioral: Dual-Task Exercise Training — Simultaneous cognitive-motor training
  Arms: Dual-Task Training

SUMMARY:
This project is focused on conducting a home-based, thinking while moving exercise intervention for adults 65 years or older, who have mild cognitive impairment, that will integrate several effective training modalities including non-contact cardio-kickboxing, stepping exercise, balance/functional training, and muscle strengthening. Cognitive function, physical function, and dual-task abilities will be assessed over the 12-week intervention and comparisons will be made between participants in the exercise intervention and control participants receiving no intervention.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Male or female
* Screened positive for mild cognitive impairment (Montreal Cognitive Assessment score 23 to 26 points
* Having no absolute contraindications to non-physician supervised exercise.

Exclusion Criteria:

* Lower-body amputation
* Non-English language speaker

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, SUNY, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from September 1st 2021 through May 21st, 2022 in local community centers, churches, and senior centers.
Groups:
- Dual-Task Training: Receives video-guided, home-based dual-task exercise
- Control: Receives no exercise guidance
Period: Overall Study
Arm/Group | Dual-Task Training | Control
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Received no exercise guidance
- Total: Total of all reporting groups
Arm/Group | Dual-Task Training | Control | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 9 | 7 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Balance: Left Limb
Description: Change in performance on the Four-Stage Balance Test: Left Limb. Minimum value: 0 seconds Maximum value: 10 seconds Higher score = better performance
Time Frame: Pre-test (time 0) and End point (12 weeks)
Population: Older adults with MCI.
Measure: Median (Inter-Quartile Range); unit: Seconds
Groups:
- Control: Control Group receives no intervention
Arm/Group | Dual-Task Training | Control
Number analyzed (Participants) | 9 | 7
Seconds | 1.52 [.78 to 2.26] | 0.05 [-0.45 to 0.55]
Statistical Analysis 1: Comparison: Dual-Task Training vs Control; Change in balance was assessed by calculating a change score between pre-test and end point scores for balance. Change scores were then compared using Mann-Whitney U test and reported as Median (Interquartile range); Test type: Superiority; p = .001, Wilcoxon (Mann-Whitney) — P-value is calculated
Statistical Analysis 2: Comparison: Dual-Task Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .003, Wilcoxon (Mann-Whitney) — P-value is calculated

2. Primary Outcome: Change in Balance: Right Limb.
Description: Change in performance on the Four-Stage Balance Test: Right Limb. Minimum value: 0 seconds Maximum value: 10 seconds Higher score = better performance
Time Frame: Pre-test (time 0) and End point (12 weeks)
Population: Older adults with MCI
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Dual-Task Training | Control
Number analyzed (Participants) | 9 | 7
seconds | 1.48 [.48 to 2.48] | 0.3 [-.30 to 0.90]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Dual-Task Training | Control
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT05108246/Prot_SAP_000.pdf